CLINICAL TRIAL: NCT02519556
Title: Randomized, Double Blind, Controlled Trial on Effectiveness Combined Probiotics in the Treatment of Atopic Dermatitis in Children
Brief Title: Trial on Effectiveness Combined Probiotics in Atopic Dermatitis in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Casa Espirita Terra de Ismael (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fabio Carmona, University of Sao Paulo, Casa Espirita Terra de Ismael
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProbioticsAD2015
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
Keywords: Probiotics; Inflammation; Awareness; Immune tolerance
MeSH Terms: conditions — Dermatitis, Atopic; Inflammation | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiatop (Experimental): Probiotic comprising the mixture of strains: Lactobacillus rhamnosus, Lactobacillus acidophilus, Lactobacillus paracasei and Bifidobacterium lactis, at a dose of 1 gram sachet, once a day for 6 months
  Interventions: Drug: Probiatop
- Placebo (Placebo Comparator): Placebo of Maltodextrin in sachet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiatop — Dilute one sachet in 100ml of water and take it in every morning, once a day for 6 months.
  Other Names: Probiotics
  Arms: Probiatop
Drug: Placebo — 1 sachet, once a day for 6 months. Dilute one sachet in 100ml of water and take it in every morning.
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
Atopic dermatitis (AD) is an immune disorder, characterized by chronic skin inflammation or relapsing, whose prevalence is increasing worldwide. Its exact etiology remains unknown. The hypothesis that an appropriate early stimulation of the intestinal flora contributes to the establishment of the immune system balance has led to the use of probiotics in the prevention and treatment of AD in several clinical and experimental studies.

Therefore, the objectives of this study will evaluate the clinical efficacy of the mixture of probiotics (Lactobacillus and Bifidobacterium) in children with AD through the SCORAD (scoring atopic dermatitis) and to evaluate the effects of this medication in the following laboratory parameters: skin prick test, total serum immunoglobulin E (IgE), inflammation composite (interferon gamma [ɣ - IFN], interleukins [IL1-β, IL-4, IL-6, IL-8] and tumor necrosis factor alpha) and immune tolerance composite (IL-10, IL-17 and transforming growth factor beta [TGF - β]).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atopic Dermatitis
* Children over 6 months.
* Teens lower than 19 years

No inclusion / Exclusion Criteria:

* Diagnostic presence or clinical signs suggesting acute or chronic skin diseases, as well as pertinent to the study, which may affect the outcome of the research.
* Being in use of drugs that can affect systemically in the course of the disease, such as systemic corticosteroids and immunosuppressants, for at least 30 days.
* Allergy or severe adverse reactions attributable to the administration of the probiotic.
* Non adherence to treatment (ie not present regular use, as prescribed) for at least one continuous month.
* Lack of attendance by more than 50% of ratings (clinical and/or laboratory) to be held during the search.
* Patient's request (or responsible's request)

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
SCORAD | 1 year
  Change from baseline in SCORAD every 3 months for 1 year

SECONDARY OUTCOMES:
Skin prick test (immediate awareness) | 1 year
Inflammation composite | 1 year
  ɣ - IFN, IL-1β, IL -4 , IL -6, IL-8 and tumor necrosis factor
Immune tolerance composite | 1 year
  IL-10, TGF - β and IL -17
Total serum IgE | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Andrade, MD, Principal Investigator — HCFMRP-USP; Persio Roxo-Junior, MD, PhD, Study Director — HCFMRP-USP; Vanessa Carregaro, PhD, Study Chair — USP-RP; Jorgete Maria e Silva, MD, Msc, Study Chair — HCFMRP-USP; Luciana Roberti, Study Chair — FMRP-USP; Laís Sacramento, Msc, Study Chair — USP-RP
Locations (1):
- Hospital das Clínicas FMRP-USP, Ribeirão Preto, São Paulo, Brazil